CLINICAL TRIAL: NCT01098604
Title: The Comparison of 32mm and 28mm Head Components in Alumina-alumina Total Hip Arthroplasty: A Randomized Clinical Trial
Brief Title: The Comparison of 32mm and 28mm Head Components in Alumina-alumina Total Hip Arthroplasty
Acronym: THA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Kyung-Hoi, Koo/professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNU 08-01
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2010-03

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 32mm ceramic head group (Active Comparator): patients performed with THA using 32mm ceramic head
  Interventions: Device: 32mm ceramic head group
- 28mm ceramic head group (Active Comparator): patients performed with THA using 28mm ceramic head
  Interventions: Device: 28mm ceramic head group

INTERVENTIONS:
Device: 32mm ceramic head group — we performed THA using 32mm ceramic head in this group.
  Arms: 32mm ceramic head group
Device: 28mm ceramic head group — we performed THA using 28mm ceramic head in this group.
  Arms: 28mm ceramic head group

SUMMARY:
It has been postulated that use of a larger femoral head could reduce the risk of dislocation after total hip arthroplasty, but only limited clinical data have been presented in third generation alumina bearings.

The purpose of this study is to evaluate the effect of femoral head size for total hip arthroplasty using third generation alumina bearings on the joint stability and clinical results.

The investigators hypothesized that larger ceramic head group has a similar rate of dislocation and clinical results in smaller ceramic head group.

ELIGIBILITY:
Inclusion Criteria:

* osteonecrosis of femoral head
* primary or secondary osteoarthritis of the hips
* femoral neck fracture

Exclusion Criteria:

* previous hemi- or total hip arthroplasty
* highly dislocated or severe ankylosed hip
* patients who are considered potentially unreliable or who may not reliably attend study visits

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
rate of dislocation in each head size | 6 weeks
  to evaluate the null hypothesis that the dislocation rate of larger ceramic head group is similar to smaller ceramic head group.
rate of dislocation in each head size | 3 months
  to evaluate the null hypothesis that the dislocation rate of larger ceramic head group is similar to smaller ceramic head group.
rate of dislocation in each head size | 6 months
  to evaluate the null hypothesis that the dislocation rate of larger ceramic head group is similar to smaller ceramic head group.
rate of dislocation in each head size | 9 months
  to evaluate the null hypothesis that the dislocation rate of larger ceramic head group is similar to smaller ceramic head group.
rate of dislocation in each head size | 12 months
  to evaluate the null hypothesis that the dislocation rate of larger ceramic head group is similar to smaller ceramic head group.
rate of dislocation in each head size | 24 months
  to evaluate the null hypothesis that the dislocation rate of larger ceramic head group is similar to smaller ceramic head group.

SECONDARY OUTCOMES:
clinical results using Harris Hip Score | 6 weeks
  to compare the clinical results such as pain, function, range of motion between both groups.
clinical results using Harris Hip Score | 3 months
  to compare the clinical results such as pain, function, range of motion between both groups.
clinical results using Harris Hip Score | 6 months
  to compare the clinical results such as pain, function, range of motion between both groups.
clinical results using Harris Hip Score | 9 months
  to compare the clinical results such as pain, function, range of motion between both groups.
clinical results using Harris Hip Score | 12 months
  to compare the clinical results such as pain, function, range of motion between both groups.
clinical results using Harris Hip Score | 24 months
  to compare the clinical results such as pain, function, range of motion between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul national University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea